CLINICAL TRIAL: NCT05728619
Title: A Phase 1b/2, Dose-finding and Expansion Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of HTMC0435 With Temozolomide in Patients With Small Cell Lung Cancer
Brief Title: HTMC0435 and Temozolomide in Treating Patients With Small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Yidian Pharmaceutical Technology Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Shanghai Huilun Pharmaceutical Co., Ltd. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HLND-01-TMZ-Ib/II-01
Record Dates: First submitted 2023-01-10; First posted 2023-02-15 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-01

CONDITIONS: Recurrent Extensive Stage Small Cell Lung Carcinoma
MeSH Terms: interventions — Temozolomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1b (Experimental): Escalating doses of HTMC0435 and Temozolomide
  Interventions: Drug: HTMC0435; Drug: Temozolomide
- Phase 2 (Experimental): Recommended phase 2 dose (RP2D) of HTMC0435 and Temozolomide
  Interventions: Drug: HTMC0435; Drug: Temozolomide

INTERVENTIONS:
Drug: HTMC0435 — Oral administration.
Drug: Temozolomide — Oral administration.

SUMMARY:
The Phase 1b part of this clinical trial is to investigate the safety and pharmacokinetic (PK) characteristics of HTMC0435 tablets combined with temozolomide in patients with various advanced solid tumors (recurrent small cell lung cancer is preferred). The Phase 2 part of the study is a multi-center, open-label, single-arm trial to investigate the preliminary efficacy of HTMC0435 and temozolomide in patients with recurrent small cell lung cancer (SCLC) at the recommended phase 2 dose.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥18 and <75 years old
2. Patients with histologically or cytologically confirmed recurrent or progressive extensive-stage SCLC, who have previously received at least first-line and no more than second-line treatments (HRR mutations are preferred)
3. [Only applicable to phase II part] At least one measurable lesion according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1)
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0~1
5. Expected survival period ≥3 months
6. Prior to the enrollment, no serious hematopoietic abnormality, and generally normal function of heart, lung, liver and kidney
7. Understand and sign the informed consent form (ICF) voluntarily. Be willing and able to complete routine visits, treatment plans, laboratory examinations and other procedures.

Exclusion Criteria:

1. Prior treatment with any poly (adenosine diphosphate [ADP]-ribose) polymerase (PARP) inhibitor
2. Prior temozolomide treatment interruption caused by toxicity
3. Received treatment with chemotherapy, radiation, biotherapy, endocrine therapy, immunotherapy, or other anti-tumor therapy ≤4 weeks prior to the first dose of HTMC0435
4. Any unrecovered AE of prior therapy ≥CTCAE 5.0 Grade 1 (except for toxicity that the investigators judged to have no safety risks, such as alopecia)
5. Currently suffering from interstitial lung disease ≥CTCAE Grade 2
6. Major surgery (excluding needle biopsy) within 4 weeks before the first dose of HTMC0435
7. Past surgical history or severe gastrointestinal diseases that the investigator believes may affect the absorption, distribution or metabolism of the study drug, such as dysphagia, active gastric ulcer, ulcerative colitis, Crohn's disease, ileus, etc.
8. History of severe cardiovascular and cerebrovascular diseases
9. Received CYP3A4 potent inhibitors or inducers within 7 days before the first dose of HTMC0435 or need to use these medications during the study
10. Symptomatic brain metastases or meningeal metastases. Patients with these metastases who have received related treatment need to meet the following conditions before they can be enrolled: no radiographic evidence of progression ≥ 4 weeks after the end of treatment; completion of treatment ≥ 28 days before the first dose; no need for systemic corticosteroids treatment (>10 mg/day prednisone or equivalent dose) within 14 days before the first dose of HTMC0435
11. Active infectious diseases which need systemic anti-infection treatment
12. Hepatitis B surface antigen (HBsAg) positive with hepatitis B virus (HBV) -DNA >1000 copies/mL or >200 IU/mL; hepatitis C virus antibody (HCV-Ab) positive
13. Human immunodeficiency virus antibody (HIV-Ab) positive
14. Previous or current diagnosis of myelodysplastic syndromes (MDS) or acute myeloid leukemia (AML)
15. Women who are pregnant or breastfeeding; women/men who are planning to have a child; women/men who refuse to use medically approved contraceptive measures for contraception during the study treatment and within 6 months after the end of the study
16. Serious psychological or mental abnormalities that may affect compliance of patients in this study
17. Current alcohol or drug abusers
18. Judgment by the investigator that the patient is not suitable for this study due to other conditions

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLT) of HTMC0435 combined with Temozolomide | Cycle 1 Day 1 to Cycle 1 Day 21
Adverse events (AE) of HTMC0435 combined with Temozolomide | Through study completion, an average of 6 months
Maximum tolerable dose (MTD) and RP2D of HTMC0435 combined with Temozolomide | Through study completion, an average of 6 months

SECONDARY OUTCOMES:
Pharmacokinetic measures - the area under the concentration-time curve from dosing (time 0) to time infinity (AUC 0-inf) | Cycle 1 Day 1 to Cycle 1 Day 9
Pharmacokinetic measures - the area under the concentration-time curve from dosing (time 0) to time t (AUC 0-t) | Cycle 1 Day 1 to Cycle 1 Day 9
Pharmacokinetic measures - apparent clearance rate (CLz/F) | Cycle 1 Day 1 to Cycle 1 Day 9
Pharmacokinetic measures - maximum plasma concentrations (Cmax) | Cycle 1 Day 1 to Cycle 1 Day 9
Pharmacokinetic measures - time to reach Cmax (Tmax) | Cycle 1 Day 1 to Cycle 1 Day 9
Pharmacokinetic measures - trough concentrations at steady state (Css, min) | Cycle 1 Day 1 to Cycle 1 Day 9
Pharmacokinetic measures - peak concentrations at steady state (Css, max) | Cycle 1 Day 1 to Cycle 1 Day 9
Pharmacokinetic measures - accumulation ratio (Rac) | Cycle 1 Day 1 to Cycle 1 Day 9
Pharmacokinetic measures - terminal plasma half-life (T1/2) | Cycle 1 Day 1 to Cycle 1 Day 9
Pharmacokinetic measures - apparent volume of distribution during terminal phase (Vz/F) | Cycle 1 Day 1 to Cycle 1 Day 9
Objective response rate (ORR) by RECIST v1.1 | Through study completion, an average of 6 months
Disease control rate (DCR) by RECIST v1.1 | Through study completion, an average of 6 months
Progression-free survival (PFS) by RECIST v1.1 | Through study completion, an average of 6 months
Duration of response (DOR) by RECIST v1.1 | Through study completion, an average of 6 months
Overall survival (OS) by RECIST v1.1 | Through study completion, an average of 6 months

OTHER OUTCOMES:
Changes in neuron-specific enolase (NSE) level from baseline | Through study completion, an average of 6 months
Changes in pro-gastrin-releasing peptide (PROGRP) level from baseline | Through study completion, an average of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yun Fan, MD, Principal Investigator — Zhejiang Cancer Hospital
Locations (3):
- China (3):
  - Zhejiang Cancer Hospital, Hangzhou
  - Jiangsu Province Hospital of Chinese Medicine, Nanjing
  - Henan Cancer Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: No